CLINICAL TRIAL: NCT03555981
Title: A Randomised Controlled Trial of Early Continuous Kangaroo Mother Care Versus Standard Care on Survival of Hospitalised Unstable Neonates <2000g in The Gambia
Brief Title: Early Kangaroo Mother Care in Gambian Hospitalised Unstable Neonates
Acronym: eKMC
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: In response to COVID pandemic
Sponsor: London School of Hygiene and Tropical Medicine (Other)
Collaborators: Wellcome Trust (Other); Medical Research Council Unit, The Gambia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14545
Record Dates: First submitted 2018-05-08; First posted 2018-06-14 (Actual); Results first posted 2023-10-16 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2019-07

CONDITIONS: Preterm Infant; Hypothermia, Newborn; Death; Kangaroo Mother Care; Infection, Bacterial
MeSH Terms: conditions — Premature Birth; Hypothermia; Death; Bacterial Infections | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Individually randomised controlled superiority trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Early KMC (Experimental): Continuous kangaroo mother care started within 24h of hospital admission, aiming for minimum 18h/day and until hospital discharge with encouragement of KMC at home
  Interventions: Other: Early Kangaroo Mother Care
- Standard care (Active Comparator): Standard care under radiant heater or incubator until clinical stability criteria are met then intermittent or continuous Kangaroo mother care started at >24h of hospital admission until hospital discharge with encouragement of KMC at home
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Early Kangaroo Mother Care — Continuous skin-to-skin contact between baby and mother/caregiver started within 24h of hospital admission
  Other Names: Early skin-to-skin contact; Early kangaroo method
  Arms: Early KMC
Other: Standard care — Incubator or radiant heater care until stable, off oxygen and >24h of admission, at which point will start intermittent or continuous kangaroo mother care
  Arms: Standard care

SUMMARY:
The mortality effect of kangaroo mother care in stable newborns <2000g is well established but mortality effect in unstable newborns is not conclusively known. This pragmatic clinical trial aims to investigate the mortality and clinical effects of early continuous Kangaroo Mother Care (KMC) compared to standard care in mild-moderately unstable neonates <2000g in a resource limited hospital setting.

DETAILED DESCRIPTION:
This individually randomised controlled trial will compare 2 parallel groups of hospitalised mild-moderately unstable neonates <2000g and aged <24h at time of screening who receive either early continuous kangaroo mother care (KMC) (started at <24h of admission) or standard care with continuous KMC at >24h of admission and when stable. The intervention will be un-blinded to participants and researchers with blinding of outcomes where possible. If participants clinically deteriorate and meet "stopping criteria" they will be temporarily withdrawn from the intervention arm and re-start KMC when clinically stable, as per the control arm. Intention to treat analysis will be used. Duration of time spent in KMC will be documented and compared between arms. All other hospital management will be provided as per a Standardised Preterm Management Protocol, based on current standard care at the study site and compliance to this protocol will be monitored in both arms.

Underlying protective mechanisms for early KMC will also be explored, focusing on causal pathways such as thermal control, cardio-respiratory stability, infection prevention control and gastro-intestinal stability pathways.

ELIGIBILITY:
Inclusion Criteria:

* New admission to study site during study period
* Admission weight <2000g
* Age 1 - 24h at start of screening
* Alive at enrolment
* Availability of study bed
* Written informed consent from parent or caregiver
* Parent or caregiver available and willing to provide intervention, if necessary

Exclusion Criteria:

* Congenital malformation incompatible with life or needing immediate surgical correction
* Severe jaundice needing immediate management
* Seizures
* Clinically stable as assessed over pre-defined period of cardio-respiratory monitoring
* Severely unstable as assessed over pre-defined period of cardio-respiratory monitoring
* Completed triplet admission
* Mother and/or neonate enrolled in another research study at time of hospital admission

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 279 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2020-04-20 (Actual); Study Completion 2020-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helen C Brotherton, MBChB, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- MRC Unit The Gambia at LSHTM, Fajara, West Coast, The Gambia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brotherton H, Gai A, Kebbeh B, Njie Y, Walker G, Muhammad AK, Darboe S, Jallow M, Ceesay B, Samateh AL, Tann CJ, Cousens S, Roca A, Lawn JE. Impact of early kangaroo mother care versus standard care on survival of mild-moderately unstable neonates <2000 grams: A randomised controlled trial. EClinicalMedicine. 2021 Aug 6;39:101050. doi: 10.1016/j.eclinm.2021.101050. eCollection 2021 Sep. PMID 34401686
- [Derived] Brotherton H, Gai A, Tann CJ, Samateh AL, Seale AC, Zaman SMA, Cousens S, Roca A, Lawn JE. Protocol for a randomised trial of early kangaroo mother care compared to standard care on survival of pre-stabilised preterm neonates in The Gambia (eKMC). Trials. 2020 Mar 6;21(1):247. doi: 10.1186/s13063-020-4149-y. PMID 32143737

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from 23rd May 2018 - 19th March 2020 at the neonatal unit of the only teaching hospital in The Gambia, providing WHO level 2+ newborn care.
Period: Overall Study
Arm/Group | Early KMC | Standard Care
Started | 138 | 141
Completed | 138 | 139
Not Completed | 0 | 2
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early KMC | Standard Care | Total
Number analyzed (Participants) | 138 | 141 | 279
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 138 | 141 | 279
  Between 18 and 65 years | NA — Neonatal trial | NA — Neonatal trial | NA — Total not calculated because data are not available (NA) in one or more arms.
  >=65 years | NA — Neonatal trial | NA — Neonatal trial | NA — Total not calculated because data are not available (NA) in one or more arms.
Age, Continuous [Median (Inter-Quartile Range); unit: hours] — hours since delivery
  hours | 2.3 [0.9 to 4.7] | 2.3 [0.7 to 5.0] | 2.3 [0.8 to 4.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 82 | 161
  Male | 59 | 59 | 118
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Gambian | 138 | 141 | 279
Region of Enrollment [Number; unit: participants]
  Gambia | 138 | 141 | 279
Admission weight [Median (Inter-Quartile Range); unit: grams] | 1459 [1204 to 1650] | 1436 [1180 to 1660] | 1450 [1180 to 1652]
Admission weight <1200g [Count of Participants; unit: Participants] | 34 | 39 | 73
Gestational age [Median (Inter-Quartile Range); unit: weeks] — Population: Gestational age data available for only 271 due to death before assessment in 8 participants
  weeks
    number analyzed (Participants) | 136 | 135 | 271
    (all) | 33 [31 to 34] | 32 [31 to 34] | 33 [31 to 34]
Twin pregnancy [Count of Participants; unit: Participants] | 41 | 45 | 86
Twin, both enrolled [Count of Participants; unit: Participants] — Twin pairs in whom both were enrolled to the trial
  Participants | 24 | 24 | 48
Stable at baseline [Count of Participants; unit: Participants] — Stable condition defined as oxygen saturation more than or equal to 88% without supplementary oxygen and with normal respiratory rate and heart rate
  Participants | 14 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: All-cause Mortality
Description: All neonatal deaths within 28 postnatal days
Time Frame: 28 days
Population: All recruited neonates with primary outcome data at 28 days were included in the analysis. This consisted of all (n=138) neonates allocated to the intervention arm and 139 neonates in the control arm, as two control participants were lost to follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Early KMC | Standard Care
Number analyzed (Participants) | 138 | 139
Participants | 29 | 34

2. Secondary Outcome: Time to Death
Description: Time from start of intervention/control procedures to death
Time Frame: 28 days of age
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Early KMC | Standard Care
Number analyzed (Participants) | 29 | 34
hours | 90.0 [65 to 172] | 98.5 [29 to 132]

3. Secondary Outcome: Cardio-respiratory Stability
Description: The 'Stability of Cardio-Respiratory in Preterm' infants is a scale to quantify the cardio-respiratory stability of preterm infants. It is composed of three parameters: Heart rate; Respiratory rate and breathing pattern and oxygen saturation (including whether is in oxygen). Scores between 0 and 2 are allocated for each parameter, with minimum total score 0 and maximum total score 6. The highest score (6) represents a better outcome, with all parameters within normal range whilst not receiving oxygen.
Time Frame: At 24 hours after start of intervention/control procedures
Population: Only neonates with outcome data available at 24h after enrolment were included in the analysis, hence the number of participants analysed is less than 279. This was principally due to mortality during first 24h of trial.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Early KMC | Standard Care
Number analyzed (Participants) | 134 | 135
units on a scale | 5 [4 to 5] | 5 [4 to 6]

4. Secondary Outcome: Number and Proportion of Participants With Hypothermia
Description: Number and proportion of participants with hypothermia (Temperature <36.5 degrees Celsius)
Time Frame: At 24 hours after start of intervention/control procedures
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Early KMC | Standard Care
Number analyzed (Participants) | 134 | 135
Participants | 51 | 55

5. Secondary Outcome: Weight Gain
Description: Average daily weight gain compared to admission weight
Time Frame: At 28 days of age
Population: Only neonates with outcome data available at age 28d were included in the analysis, hence the number of participants analysed is less than 279. This was principally due to mortality, loss to follow up and small number of participants with missing data
Measure: Mean (Standard Deviation); unit: grams/day
Arm/Group | Early KMC | Standard Care
Number analyzed (Participants) | 103 | 101
grams/day | 10.3 (10.1) | 12.5 (12.1)

6. Secondary Outcome: Exclusive Breastfeeding
Description: Number of babies who are exclusively breastfed (defined as only receiving breast milk with no infant formula supplementation)
Time Frame: At time of hospital discharge, within study period, on average 2 weeks of age
Population: Only neonates with outcome data available at discharge were included in the analysis, hence the number of participants analysed is less than 279. The missing data was principally due to mortality prior to discharge.
Measure: Count of Participants; unit: Participants
Arm/Group | Early KMC | Standard Care
Number analyzed (Participants) | 109 | 107
Participants | 107 | 105

7. Secondary Outcome: Suspected Infection Between 3d to 28d of Age
Description: Number and proportion of participants with suspected infection between 3d to 28d of age, or age at latest follow up
Time Frame: Within 28 days of age
Population: All randomised participants were included in the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Early KMC | Standard Care
Number analyzed (Participants) | 138 | 141
Participants | 28 | 21

8. Secondary Outcome: Neonatal Intestinal Carriage of Extended Spectrum Beta-Lactamase-producing Klebsiella Pneumoniae
Description: Number and proportion of participants with intestinal carriage of Extended Spectrum Beta-Lactamase-Klebsiella pneumoniae
Time Frame: At day 28 of age
Reporting Status: Not Posted, anticipated posting 2024-04

9. Secondary Outcome: Duration of Hospital Admission
Description: Mean length of admission (first admission only if re-admitted)
Time Frame: Within 28 days of age or at latest follow-up
Population: Only neonates with outcome data available at time of discharge were included in the analysis, hence the number of participants analysed is less than 279. Neonates were died during first hospital admission were not included in the analysis.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Early KMC | Standard Care
Number analyzed (Participants) | 103 | 101
Days | 16.6 (11.1) | 16.3 (10.0)

ADVERSE EVENTS:
Time Frame: 28 postnatal days
Description: Only serious adverse events were monitored/assessed. Other adverse events were not monitored/assessed.
Arm/Group | Early KMC | Standard Care
All-Cause Mortality (participants affected / at risk) | 29/138 | 34/141
Serious Adverse Events (participants affected / at risk) | 30/138 | 28/141
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Early KMC (N=138) | Standard Care (N=141)
Life threatening event (General disorders) | 13 (13) | 11 (11) — Defined as either apnoea needing resuscitation, severe instability as per protocol definitions or any other life threatening event as assessed by a clinician
Risk of disability (Nervous system disorders) | 6 (6) | 7 (7) — Any condition placing the neonate at increased risk of permanent or temporary disability, such as suspected meningitis, severe jaundice or acquired hydrocephalus
Hospital re-admission (General disorders) | 4 (4) | 5 (5) — Re-admission within 28 postnatal days
Prolonged hospitalisation (General disorders) | 7 (7) | 5 (5) — Hospitalised for >28 days

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-03-18): https://cdn.clinicaltrials.gov/large-docs/81/NCT03555981/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-24): https://cdn.clinicaltrials.gov/large-docs/81/NCT03555981/SAP_001.pdf